CLINICAL TRIAL: NCT00015249
Title: Prepulse Inhibition of Startle in Cocaine Dependence (Human)
Brief Title: Prepulse Inhibition of Startle in Cocaine Dependence - 7
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: New York MDRU (Other)
Masking: Double | Purpose: Diagnostic
Other Study IDs: NIDA-5-0013-7; Y01-5-0013-7
Record Dates: First submitted 2001-04-18; First posted 2001-04-18 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1998-06

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Amantadine

INTERVENTIONS:
Drug: Amantadine

SUMMARY:
The purpose of this study is to assess the effects of chronic cocaine use on the acoustic startle response and on gating of this response in humans.

DETAILED DESCRIPTION:
The objective of this study is to assess the effects of chronic cocaine use on the acoustic startle response and on gating of this response in humans.

ELIGIBILITY:
Inclusion Criteria:

Cocaine dependence. Male. Right handed. Negative urine for cocaine

Exclusion Criteria:

Positive urine for cocaine. History of head trauma. Significant medical disease.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1997-02; Primary Completion 1998-04 (Actual); Study Completion 1998-05 (Actual)

PRIMARY OUTCOMES:
Percent prepulse inhibition
Cocaine assessment

CONTACTS AND LOCATIONS:
Overall Officials: John Rotrosen, M.D., Principal Investigator — New York MDRU
Locations (1):
- New York MDRU, New York, New York, United States

REFERENCES:
- [Background] CPDD, 98, 99 NIDA Research Monograph Series 179, 1998 Manuscript submitted..